CLINICAL TRIAL: NCT04943510
Title: Characterization of Hamstring and Quadriceps Neuromuscular Fatigue After Different Modality of Training in Soccer Players
Brief Title: Characterization of Hamstring and Quadriceps Neuromuscular Fatigue After Soccer Game
Acronym: QIF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8168
Record Dates: First submitted 2021-06-02; First posted 2021-06-29 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Neuromuscular Fatigue; Exercise
Keywords: Hamstring; Neuromuscular fatigue; Soccer; Performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: three randomizations will be used to determine the order of the tests that will be proposed to the subjects:
  * on the one hand for the exercise modalities (match, anaerobic, aerobic)
  * and, on the other hand, for the exercise modalities included in the anaerobic and aerobic exercise families: Anaerobic agility / anaerobic - linear sprints Aerobic - shuttle / aerobic - linear
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical exercices arm (Experimental): three randomizations will be used to determine the order of the tests that will be proposed to the subjects: on the one hand for the exercise modalities (match, anaerobic, aerobic) and, on the other hand, for the exercise modalities included in the anaerobic and aerobic exercise families: Anaerobic agility / anaerobic - linear sprints Aerobic - shuttle / aerobic - linear
  Interventions: Other: Physical exercices

INTERVENTIONS:
Other: Physical exercices — surface EMG: surface electrodes will be positioned on the muscles to evaluate the level of muscle activation
  non invasive muscular neurostimulations : application of a percutaneous electrical stimulation of the motor nerve of the considered muscle and a direct electrical stimulation of the muscle
  Other Names: Non invasive muscular neurostimulations; Surface EMG

SUMMARY:
This is a monocentric study comparing hamstring and quadriceps neuromuscular fatigue after simulated soccer game, anaerobic and aerobic training sessions. The purpose of this study was:

1. To quantify the decrease of isometric force immediately after a simulate soccer game.
2. To characterize peripheral and central fatigue between hamstring and quadriceps muscles and described the kinetics of recovery after specific tasks of soccer training.
3. To compare the level neuromuscular fatigue induced by anaerobic and aerobic training.
4. To highlight correlation between neuromuscular fatigue and performance markers.

ELIGIBILITY:
Inclusion Criteria:

* male
* age limits: minimum: 16 ; maximum: 40 years old
* to be a soccer player, licensed to the French Football Federation
* affiliation to the social health insurance scheme
* signing an informed consent form

Exclusion Criteria:

* impossibility to give the subject enlightened information (subject in emergency situation, difficulties in understanding the study, …)
* subject under the protection of justice
* subject under guardianship or curatorship
* lower limbs musculotendinous or articular problems
* smoker or having been a smoker in the last 5 years
* subject wearing a pacemaker
* drug treatment in progress and impossibility to stop it within 7 days before the beginning of the study.

Ages: 16 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Difference in maximal isometric hamstring strength before and immediately after exercise (i.e., pre vs. immediate post exercise) expressed as a percentage (%). | Before and immediately post exercise (i.e., during the first minute after cessation of exercise)

SECONDARY OUTCOMES:
Relative difference (in %) in maximum isometric hamstring strength before and after exercise (i.e., pre- vs. post-exercise), relative to pre-exercise strength across different test types. | Before and immediately post exercise, 5, 10, 15, 30-minutes and 24 and 48-hours post-exercise
Relative difference (in %) in maximal isometric quadriceps strength before and after exercise (i.e., pre vs. post exercise), related to preexercise strength according to the different types of tests. | Before and immediately post exercise, 5, 10, 15, 30-minutes and 24 and 48-hours post-exercise
Relative difference (%) in maximum isometric hamstring and quadriceps strength for each test type at the different times of interest. | Before and immediately post exercise, 5, 10, 15, 30-minutes and 24 and 48-hours post-exercise
Difference in pre- and post-exercise (i.e., pre- vs. post-exercise) hamstring potentiated jerk amplitude (N) relative to pre-exercise amplitude by event type at different times of interest. | Before and immediately post exercise, 5, 10, 15, 30-minutes and 24 and 48-hours post-exercise
Difference in pre- and post-exercise (i.e., pre- vs. post-exercise) potentiated jerk amplitude (N) of the quadriceps, relative to pre-exercise amplitude, by test type at different times of interest. | Before and immediately post exercise, 5, 10, 15, 30-minutes and 24 and 48-hours post-exercise
Difference in amplitude of the potentiated jerk (N) before and after exercise, related to the preexercise amplitude according to the muscle involved (hamstrings or quadriceps) and the type of test at different times of interest. | Before and immediately post exercise, 5, 10, 15, 30-minutes and 24 and 48-hours post-exercise
Difference in the level of voluntary hamstring activation, expressed in newtons (N), before and after exercise, related to the pre-exercise action level, according to the type of test at different times of interest. | Before and immediately post exercise, 5, 10, 15, 30-minutes and 24 and 48-hours post-exercise
Difference in the level of voluntary quadriceps activation, expressed in newtons (N), before and after exercise, related to the pre-exercise action level, according to the type of test at different times of interest. | Before and immediately post exercise, 5, 10, 15, 30-minutes and 24 and 48-hours post-exercise
Difference in the level of voluntary action before and after exercise, related to the level of action before exercise, according to the muscle involved (hamstrings or quadriceps) and the type of test at different times of interest. | Before and immediately post exercise, 5, 10, 15, 30-minutes and 24 and 48-hours post-exercise
Differences in overall fatigue, peripheral fatigue, and central fatigue of hamstrings versus quadriceps between exercise modalities. | Before and immediately post exercise, 5, 10, 15, 30-minutes and 24 and 48-hours post-exercise
  Determine the modalities of exercises which induce the highest level of fatigue and characterize the etiology of neuromuscular fatigue (i.e., peripheral or central) for typical drills performed daily by elite soccer players
Ratio (%) of initial to post-exercise values based on field indicators and neuromuscular fatigue. | Before and immediately post exercise, 5, 10, 15, 30-minutes and 24 and 48-hours post-exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Universitaires de Strasbourg, Strasbourg, France